CLINICAL TRIAL: NCT00197132
Title: A Single-centre, Randomised, Double-blind, Placebo Controlled, Two 12 Week Period, Cross-over Phase III Study to Investigate the Effect of Rosiglitazone 4mg bd on the Vasodilator Response to Hyperinsulinaemia in Obese Insulin Resistant Subjects.
Brief Title: Study In Patients With Insulin Resistance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 49653/375
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Insulin Resistance
Keywords: Insulin resistance vasodilatory response
MeSH Terms: conditions — Insulin Resistance | interventions — Rosiglitazone

INTERVENTIONS:
Drug: Avandia

SUMMARY:
Fluid management study in patients with insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-36 kg/m2 inclusive and at least two additional features of the metabolic syndrome or a first degree relative with a history of type 2 diabetes mellitus. BMI = Weight/height², (where weight is in kg, height in m).
* Male or female aged 30 to 65 years, inclusive, at screening.
* Female subjects must be post-menopausal (i.e. >6 months without menstrual period), surgically sterile, or using effective contraceptive measures (oral contraceptives, Norplant Depo-Provera) or intra-uterine devices (IUD) (a diaphragm with spermicide or a condom with spermicide). Women of childbearing potential must use effective contraceptive measures for at least 1 month prior to visit 1, and should continue to use the same contraceptive method during the study and for 30 days after discontinuing study treatment.
* Willing and able to provide a signed and dated written informed consent.

Exclusion Criteria:

* Subjects with type 2 diabetes mellitus defined as an HbA1c level >6.5% or a fasting plasma glucose of > 7.0 mmol/L. If fasting plasma glucose is between 6.1 and 7.0 mmol/L then a 75 g oral glucose test will be performed to exclude diabetes mellitus.
* Subjects who have initiated lipid lowering therapy within the last 6 months and subjects who have increased the dose of these therapies within the last 3 months prior to study start.
* Subjects who are taking Non Steroidal Anti-inflammatory Drugs, fibrates, anticoagulants or cardiovascular medications (β-blockers, nitrates, calcium antagonists, ACE inhibitors, angiotensin II antagonists, alpha blockers, diuretics, centrally acting anti-hypertensives, directly acting antihypertensives e.g., diazoxide, digoxin, anti-arrhythmics) and are unable to stop these medications for the duration of the study.
* Exposure to a thiazolidinedione (TZD) or other PPAR-γ agonist (e.g. rosiglitazone, troglitazone, pioglitazone, G1262570) within the last 4 months or participation in a clinical study involving a TZD or PPAR-γ agonist.
* Subjects who have required the use of any anti-diabetic medication at any time.
* Use of any investigational drug within 30 days preceding the first dose of medication at the start of the study.
* Subjects with a documented history of significant hypersensitivity (e.g. difficulty swallowing, difficulty breathing, tachycardia or skin reaction) to thiazolidinediones or PPAR-γ agonists.
* Systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg or receiving antihypertensive therapy.
* Subjects with unstable or severe angina (requiring continual therapy) or congestive heart failure.
* Presence of clinically significant hepatic disease.
* Clinically significant anaemia.
* Subjects with creatinine clearance <40 mL/min.
* Women who are lactating, pregnant or planning to become pregnant during the course of the study.
* Alcohol or drug abuse within the last 6 months.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-10; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow

SECONDARY OUTCOMES:
Insulin sensitivity, plasma volume, transcapillary escape rate, inhibition to vasodialtory response, changes in cardiac output, plasma catecholamine levels, changes in plasma hormone/markers of vascular permeability, safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 49653/375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 49653/375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 49653/375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 49653/375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 49653/375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 49653/375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 49653/375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register